CLINICAL TRIAL: NCT05170022
Title: Clinical Profile in Patients With Essential Tremors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zozil yousef zakaria, principal investigator, Assiut University
Other Study IDs: essential tremors
Record Dates: First submitted 2021-12-10; First posted 2021-12-27 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Essential tremors are no longer a single motor disorder but disorder of movement associated with non-motor symptoms and the aim of this study is to explore the clinical profile of patients with essential tremors including motor and non-motor features and their relationship.

and to identify clinical predictors of these features.

DETAILED DESCRIPTION:
Essential tremors (ET) was defined as mono-symptomatic tremor syndrome involving both upper limbs during action for at least 3 years, with or without tremor in other body parts . ET is considered the most prevalent adult movement disorder, The crude prevalence of ET varies widely from 0.08 to 220 cases per 1000 persons. Many pathological post-Mortem studies are providing evidence that ET is mostly can be recognizes as neurodegenerative disease of the cerebellum and brain stem .

In the last decade there is an emerging studies that discuss the presence of associated motor, non- motor, sensory and psychological symptoms besides the tremors . Motor features of ET are not confined to tremors. Another feature of ET is gait ataxia , Eye movement abnormalities of subclinical degree, difficulties in learning motor skills, Bradykinesia and slowness of finger tapping .

Studies of the last two decades reported mild cognitive deficits in patients with ET in comparison to healthy controls. These deficits affect number of cognitive domains, especially verbal memory, naming, verbal fluency, attention- concentration, working memory and concept formation . In addition ET was found to be associated with hearing impairment with abnormal threshold at higher tone frequencies which refer to sensorineural hearing loss, and olfactory deficits which both may points to cochlear pathology. Moreover, patients with ET thought to have higher incidence of depression and anxiety symptoms than age-matched healthy individuals correlated with tremors severity .

ELIGIBILITY:
Inclusion Criteria:

1. All adults Patients are fulfilling cases definition of essential tremors will be included.
2. Gender: both sexes are included.
3. Any patient is, able to provide informed consent including permission to obtain information from patients' clinical medical history of at least three years' duration

Exclusion Criteria:

1. Patients are diagnosed with other neurological disorders unrelated to essential tremors.
2. Patients had any other condition presented with other cognitive or psychiatric disorders or known as drug abusers.
3. Patient had any systemic disease presented with tremors rather than essential tremors or compliant on medication had tremors side effect.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All cases are recruited in the study period; six months duration since date of approval of ethical committee of Assiut University hospitals and postgraduate committee of Faculty of Medicine, Assiut University.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Determine clinical profile including motor and non-motor features in these patients | 3 years
  describing the motor and non-motor associations ( cognitive , psychological and sensory )with essential tremors.

SECONDARY OUTCOMES:
To identify clinical predictors of these features. | 3 years
  Determine the clinical predictors for these features in these ET patients and impact on their quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Abo-lftoh, prof. doctor, Study Director — hospital medical school affiliation; Nourelhoda Ah Haridy, doctor, Study Director — hospital medical school affiliation
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Elbelkemy M, Shalash A, Mansour A, Hamed E, Abdelalim HM. Non motor symptoms in patients with essential tremor. QJM An Int J Med. 2020;113(Supplement_1):1-4.
- [Background] Bhatia KP, Bain P, Bajaj N, Elble RJ, Hallett M, Louis ED, Raethjen J, Stamelou M, Testa CM, Deuschl G; Tremor Task Force of the International Parkinson and Movement Disorder Society. Consensus Statement on the classification of tremors. from the task force on tremor of the International Parkinson and Movement Disorder Society. Mov Disord. 2018 Jan;33(1):75-87. doi: 10.1002/mds.27121. Epub 2017 Nov 30. PMID 29193359
- [Background] Huang H, Yang X, Zhao Q, Ning P, Shen Q, Wang H, Xie D, Lu H, Xu Y. Clinical characteristics of patients with essential tremor or essential tremor plus. Acta Neurol Scand. 2020 Apr;141(4):335-341. doi: 10.1111/ane.13209. Epub 2020 Jan 6. PMID 31863462
- [Background] Rao AK, Louis ED. Ataxic Gait in Essential Tremor: A Disease-Associated Feature? Tremor Other Hyperkinet Mov (N Y). 2019 Jun 19;9. doi: 10.7916/d8-28jq-8t52. eCollection 2019. PMID 31413894
- [Background] Gitchel GT, Wetzel PA, Baron MS. Slowed saccades and increased square wave jerks in essential tremor. Tremor Other Hyperkinet Mov (N Y). 2013 Sep 3;3:tre-03-178-4116-2. doi: 10.7916/D8251GXN. eCollection 2013. PMID 24116343
- [Background] Shill HA, De La Vega FJ, Samanta J, Stacy M. Motor learning in essential tremor. Mov Disord. 2009 Apr 30;24(6):926-8. doi: 10.1002/mds.22479. PMID 19243062
- [Background] Bologna M, Paparella G, Colella D, Cannavacciuolo A, Angelini L, Alunni-Fegatelli D, Guerra A, Berardelli A. Is there evidence of bradykinesia in essential tremor? Eur J Neurol. 2020 Aug;27(8):1501-1509. doi: 10.1111/ene.14312. Epub 2020 May 31. PMID 32396976
- [Background] Louis ED, Joyce JL, Cosentino S. Mind the gaps: What we don't know about cognitive impairment in essential tremor. Parkinsonism Relat Disord. 2019 Jun;63:10-19. doi: 10.1016/j.parkreldis.2019.02.038. Epub 2019 Mar 1. PMID 30876840
- [Background] Bermejo-Pareja F, Puertas-Martin V. Cognitive features of essential tremor: a review of the clinical aspects and possible mechanistic underpinnings. Tremor Other Hyperkinet Mov (N Y). 2012;2:02-74-541-1. doi: 10.7916/D89W0D7W. Epub 2012 Sep 14. PMID 23440004
- [Background] Yilmaz NH, Akbostanci MC, Yilmaz N. Sensorineural Hearing Loss in Non-depressed Essential Tremor Cases and Controls: A Clinical and Audiometric Study. Tremor Other Hyperkinet Mov (N Y). 2015 Jan 29;5:281. doi: 10.7916/D8XW4HKQ. eCollection 2015. PMID 25667817
- [Background] Shalash AS, Mohamed H, Mansour AH, Elkady A, Elrassas H, Hamid E, Elbalkimy MH. Clinical Profile of Non-Motor Symptoms in Patients with Essential Tremor: Impact on Quality of Life and Age-Related Differences. Tremor Other Hyperkinet Mov (N Y). 2019 Dec 6;9. doi: 10.7916/tohm.v0.736. eCollection 2019. PMID 31867132
- [Background] Rahman TT, El Gaafary MM. Montreal Cognitive Assessment Arabic version: reliability and validity prevalence of mild cognitive impairment among elderly attending geriatric clubs in Cairo. Geriatr Gerontol Int. 2009 Mar;9(1):54-61. doi: 10.1111/j.1447-0594.2008.00509.x. PMID 19260980
- [Background] Wechsler memory scale. - PsycNET [Internet]. [cited 2021 Oct 25]. Available from: https://psycnet.apa.org/record/1946-00348-000
- [Background] 36-Item Short Form Survey (SF-36) Scoring Instructions | RAND [Internet]. [cited 2021 Oct 23]. Available from: https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/scoring.html
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] HAMILTON M. The assessment of anxiety states by rating. Br J Med Psychol. 1959;32(1):50-5. doi: 10.1111/j.2044-8341.1959.tb00467.x. No abstract available. PMID 13638508
- [Background] Williams JB. A structured interview guide for the Hamilton Depression Rating Scale. Arch Gen Psychiatry. 1988 Aug;45(8):742-7. doi: 10.1001/archpsyc.1988.01800320058007. PMID 3395203
- [Background] Shill HA, Adler CH, Sabbagh MN, Connor DJ, Caviness JN, Hentz JG, Beach TG. Pathologic findings in prospectively ascertained essential tremor subjects. Neurology. 2008 Apr 15;70(16 Pt 2):1452-5. doi: 10.1212/01.wnl.0000310425.76205.02. PMID 18413570